CLINICAL TRIAL: NCT01883674
Title: Milk and Milk-produce to Counteract the Loss of Muscle Mass and Function in Exercising Older Adults.
Acronym: PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLC-021742
Record Dates: First submitted 2013-02-07; First posted 2013-06-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Physical capacity; Muscle force; Muscle quality; Milk proteins; Essential amino acids; Proteins; Resistance training; Exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Milk proteins (Experimental): This group will do a resistance training + milk proteins (milk beverage)
  Interventions: Other: Resistance training
- Essential amino acids (add to soya bvg) (Experimental): This group will do a resistance training + essential amino acids (added to soya beverage)
  Interventions: Other: Resistance training
- No protein (control) (Placebo Comparator): This group will do a resistance training + ingestion of the control beverage (no protein, rice beverage)
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — All group will exercise 3x/week. Each session of resistance training will last 60min. and will target main muscular groups.

SUMMARY:
This project evaluates the use of different types of proteins from various food sources after an exercise session, on muscle mass and physical capacity in aged sarcopenic men (who have low muscle mass). Specifically, researchers want to:

* Examine the efficiency of protein intake after exercise on muscle mass and physical abilities;
* Examine the impact of exercise and proteins on blood lipids (LDL cholesterol, HDL cholesterol, total cholesterol and triglycerides);
* Examine the impact of exercise and proteins on liver enzymes;
* Examine the impact of exercise and proteins on a hormone that controls hunger;
* Evaluate the program's impact on the ability of the body to produce energy.

All participants are exercising (resistance training) and ingest one of the 3 different sources of proteins, immediately after training:

* Milk proteins (from milk beverage)
* Essential amino acids (added to a soya beverage)
* No protein (rice beverage - control group)

Our hypothesis is that proteins from milk will induce a gain in muscle mass and physical function equivalent to the essential amino acids (EAA). We anticipate that both milk proteins and EAA will be both superior to control group.

This would represent an interesting finding since milk is more accessible, palatable and cheaper than essential amino acids commercial mix.

ELIGIBILITY:
Inclusion Criteria:

* 65-75 years
* francophone or understanding French
* muscle mass index < 10.75 kg/m2 (Janssen et al, 2004)
* body mass index <30kg/m²
* weight stable (< 2 kg) for 6 mo
* no resistance exercise for 3 years
* controlled blood pressure for at least 6 months

Exclusion Criteria:

* major physical disability
* medical treatment influencing metabolism
* statin treatment
* diagnosis or any sign of kidney disease

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Muscle mass | At baseline and post intervention (17th week)

SECONDARY OUTCOMES:
Relative strength | At baseline and post intervention (17th week)
Blood markers of inflammation | At baseline and post intervention (17th week)
  Plasmatic IL-6 anf TNF-alpha
Plasma Lipid profile | At baseline and post intervention (17th week)
  Apolipoproteins (Apo-AI, Apo-AII, Apo-B); Total cholesterol, HDL, LDL and triglycerides.
Plasma creatinine | At baseline, mid (8th week) and post intervention (17th week)
  Blood marker on renal function will be assessed to ensure the safety of the supplementation of protein intake on renal function in sarcopenic men.
Blood markers of fatty liver | At baseline and post intervention (17th week)
  Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Gamma-glutamyltransferase (GGT) and Alkaline phosphatase (ALP).
extracellular HSP72 | At baseline and post intervention (17th week)

OTHER OUTCOMES:
Dietary intakes | At baseline, mid (8th week) and post intervention (17th week)
  3-day food record - Control variable (in order to verify if changes we observe through the intervention are accountable or not for dietary intakes)
Physical activity level | At baseline and post intervention (17th week)
  Physical Activity Scale for the Elderly (PASE) - Control variable (in order to verify if changes we observe through the intervention are accountable or not for daily physical activity level)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle J. Dionne, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le vieillissement, Sherbrooke, Quebec, Canada